CLINICAL TRIAL: NCT01677598
Title: A Study to Evaluate Ustekinumab in Clinical Practice in Patients With Plaque Psoriasis in Asia-Pacific Countries
Brief Title: A Study to Evaluate Ustekinumab in Patients With Plaque Psoriasis in Asia-Pacific Countries
Acronym: MARCOPOLO
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100140; CNTO1275PSO4016 (Other: Johnson & Johnson Pte Ltd)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Ustekinumab; CNTO 1275; Asia-Pacific
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Patients with plaque psoriasis: Patients with plaque psoriasis using ustekinumab in Asia-Pacific countries.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — No intervention will be administered during study. This will be an observational study in patients using ustekinumab as label-recommended or other/missed dose interval in Asia-Pacific countries
  Other Names: CNTO 1275

SUMMARY:
The purpose of this study is to determine how patients use ustekinumab (label-recommended or other/missed dose interval) in Asia-Pacific countries.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the medication), multicenter, Phase 4, observational study (no study medication was administered during the study) designed to assess how patients will use ustekinumab (label-recommended or other/missed dose interval) in Asia-Pacific countries. The study will consist of 4 study visits which will take place over the duration of 1 year. At the first visit (ie, Week 0), eligibility for the study will be determined (it will be screening and baseline visit). At each subsequent visit (Weeks 16, 28, and 52), exposure to ustekinumab will be recorded, questionnaires for efficacy will be completed, and information about adverse events and concomitant medications will be collected. As many patient reported outcome questionnaires as possible will be administered, depending on the availability of validated translations. Safety will be assessed by monitoring of adverse events, vital signs and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque psoriasis, according to the dermatologists' clinical judgment
* Agree to initiate treatment with ustekinumab on the same day as enrollment into the study
* Have not received anti-IL12/23 therapies within 6 months prior to enrollment into the study

Exclusion Criteria:

* Has difficulty understanding questions posed by any of the questionnaires
* Are currently participating in an investigational drug clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years of age with a diagnosis of plaque psoriasis, according to the dermatologists' clinical judgment
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2011-12-02 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
Number of psoriasis patients who use ustekinumab with label-recommended interval or other/missed dose interval | up to 52 weeks
  Number of psoriasis patients who use ustekinumab with label-recommended interval or other/missed dose interval will be assessed at Weeks 0, 16, 28, 52.

SECONDARY OUTCOMES:
Epidemiologic characteristics of the psoriasis population | Week 0
  Epidemiologic characteristics of the psoriasis patients (sex, age, race, weight height, and peak disease level) will be determined.
Change from baseline (Week 0) in Psoriasis Area and Severity Index (PASI) score at Weeks 16, 28 and 52 | Baseline (Week 0), Weeks 16, 28 and 52
  The PASI is a physician-administered assessment tool used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease).
Change from baseline (Week 0) in Nail Psoriasis Severity Index (NAPSI) score at Weeks 16, 28, and 52 | Baseline, Weeks 16, 28 and 52
  NAPSI is used for assessing and grading the severity of nail psoriasis. Each nail is divided with imaginary horizontal and longitudinal lines into quadrants. Each nail is given a score for nail matrix psoriasis (0 to 4) and nail bed psoriasis (0 to 4) depending on the presence of any of the features of nail psoriasis in the 4 quadrants as: 0 (none), 1 (present in 1/4 nail), 2 (2/4), 3 (3/4), and 4 (4/4). Each nail gets a matrix score and a nail bed score, the total of which is the score for that nail (0 to 8). Each nail is evaluated, and the sum of all the nails is the total NAPSI score. The sum of the scores from all nails is 0 to 160 (Both finger and toe nails are included). Higher scores indicate worsening.
Change from baseline in EuroQol 5 Dimensional Questionnaire (EQ-5D) index score and EQ visual analog scale (VAS) at Weeks 16, 28, and 52 | Baseline, Weeks 16, 28 and 52
  The EQ-5D (EuroQol Group) is a validated generic measure of quality of life which usually requires less than 1 minute to complete (eg, the questionnaire may have questions about mobility, self care, usual activities, pain/discomfort and anxiety/depression.
Change from baseline (Week 0) in Dermatology Life Quality Index (DLQI) score | Baseline, Weeks 16, 28 and 52
  The DLQI is a patient-completed 10-item questionnaire that, in addition to evaluating overall quality of life, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The aim of this questionnaire is to measure how much your skin problem has affected your life over the last week. For each of 10 questions patient has to select one of the following options: very much, a lot, a little, not at all.
Change from baseline (Week 0) in Patient Benefit Index (PBI) score at Weeks 16, 28, and 52 | Baseline, Weeks 16, 28 and 52
  The PBI is a patient-defined benefit assessment tool. Patients select personally relevant treatment goals from a standardized list of benefits called the Patient Needs Questionnaire. An evaluation of those treatment goals assessed by the patient is captured on the Patient Benefit Questionnaire. The PBI is calculated from the sum of the benefit items weighted by their respective relevance divided by the number of relevant items. Values between 0 (no benefit) and 4 (maximal patient-defined benefit) are possible.
Number of patients achieving PASI 50, 75, and 90 response (ie, at least 50%, 75% and 90% improvement in PASI) | up to 52 weeks
  Number of patients achieving PASI 50, 75, and 90 response (ie, at least 50%, 75% and 90% improvement in PASI) will be evaluated at Weeks 16, 28, and 52.
Number of patients achieving a DLQI improvement (reduction) of greater than or equal to 5 points | up to 52 weeks
  Number of patients achieving a DLQI improvement (reduction) of greater than or equal to 5 points will be evaluated at Weeks 16, 28, and 52.
Number of patients achieving a score of 0 or 1 in DLQI | up to 52 weeks
  Number of patients achieving a score of 0 or 1 in DLQI will be evaluated at Weeks 16, 28, and 52.
Number of patients achieving an improvement in PBI | up to 52 weeks
  Number of patients achieving an improvement in PBI will be evaluated at Weeks 16, 28, and 52.
Number of patients with comorbidities (obesity, hypertension, diabetes, dyslipidemia, and heart disease) | up to 52 weeks
  Number of patients with comorbidities (obesity, hypertension, diabetes, dyslipidemia, and heart disease) will be evaluated at baseline, Weeks 16, 28, and 52.
Health Economics/Medical Resource Utilization Questionnaire (HE/MRU) | up to 52 weeks
  Health economic impact using the HE/MRU questionnaire will be assessed at baseline, Weeks 16, 28 and 52. Patients will be asked to complete a HE/MRU questionnaire to collect information on demographics, medical insurances, and use of biologic agents and phototherapy. Sections 1 and 2 are completed by the patient. Sections 3 and 4 are completed by the physician.
Change from baseline in productivity VAS at Weeks 16, 28, and 52 | Baseline, Weeks 16, 28 and 52
  A 10 cm VAS will be used to assess work, school, or at home productivity. Patients will be asked to put a single vertical line across the horizontal line at the spot that they feel best reflects the answer to the question, "How much has your disease affected your daily productivity at work, school or at home in the past 4 weeks?" The score will be recorded as a measurement of the placement of the patient's mark on a 10 cm scale.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- Jakarta Pusat, Indonesia
- Malaysia (2):
  - Johor Bahru
  - Pulau Pinang
- Singapore, Singapore
- South Korea (4):
  - Incheon
  - Seongnam-Si, Gyeonggi-Do
  - Seoul
  - Suwon
- Taipei, Taiwan